CLINICAL TRIAL: NCT05599854
Title: Short-term Anterior Segment Changes After Pars Plana Vitrectomy (PPV) and Silicone Oil (SO) Tamponade, Anterior Segment OCT (AS-OCT) Study.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sarah Alaa Ezzat Abdelmoneim, Dr., Assiut University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Screening
Other Study IDs: ASOCT changes after vitrectomy
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: ASOCT Changes After Vitrectomy and Silicone Oil Injection
Keywords: ASOCT, vitrectomy, silicone oil injection
MeSH Terms: interventions — Vitrectomy; Silicone Oils; Predictive Value of Tests; styrene-oxide isomerase

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: vitrectomy and silicone oil injection — Parsplana vitrectomy and silicone oil injection
  Other Names: PPV and SOI

SUMMARY:
The purpose of our study is to utilize AS-OCT to analyze the anterior segment morphological changes in the early postoperative period of patients who will undergo PPV with silicone oil injection.

DETAILED DESCRIPTION:
1. Type of the study: A prospective comparative study.
2. Study Setting: Assiut university hospital.
3. Study subjects:

   1. Inclusion criteria:

      Patients suffering from different vitreo-retinal disorders (rhegmatogenous retinal detachment, diabetic vitreous hemorrhage, diabetic tractional retinal detachment) with either preserved crystalline lens or previous cataract surgery (at least 3 months prior to PPV) will be recruited
   2. Exclusion criteria:

      Patient with previous history of ocular trauma, co-existing glaucoma, co-existing anterior uveitis, complicated cataract surgery, IOL-related complications, previous vitreo-retinal surgery, visually significant cataract (necessitating combined phacoemulsification with PPV and SO) and significant corneal opacity will be excluded. If any significant post-PPV complication develops, patient will be excluded from the study.
   3. Sample Size Calculation:

      Thirty eyes (30 patients) will undergo PPV with SO tamponade and AS-OCT analysis prior to surgery and 1 week post-operatively to achieve study power of 80% with 0.05 significance.

      4 -Study tools (in detail, e.g., lab methods, instruments, steps, chemicals, …): All participants underwent best-corrected visual acuity (BCVA) by Snellen's chart, Slit lamp assessment of the anterior segment, dilated fundus examination, intra-ocular pressure (IOP) measurement by calibrated Goldmann Applanation Tonometer (GAT). Baseline Ophthalmic ultrasound and Axial length measurement will be obtained.

      Anterior segment OCT (AS-OCT) protocol All eyes will be examined by AS-OCT (Nidek RS-3000 Advance, Tokyo, Japan) 1-2 days prior to vitreo-retinal surgery and one week after surgery by single experienced physician. Poor fixation or poor image signal (less than 3/10) will exclude the patient from the study.

      Anterior segment OCT (AS-OCT) parameters The following anterior segment parameters will be evaluated; central and peripheral anterior chamber depth (cACD, pACD), anterior chamber angle (ACA) and central corneal thickness (CCT).

      5 -Research outcome measures:

   <!-- -->

   1. Primary (main):

      Mean change in central anterior chamber depth after PPV with SO tamponade.
   2. Secondary (subsidiary):

Mean change in peripheral anterior chamber depth, mean change in anterior chamber angle and mean change anterior chamber angle entry area.

ELIGIBILITY:
Inclusion Criteria:

Patients suffering from different vitreo-retinal disorders (rhegmatogenous retinal detachment, diabetic vitreous hemorrhage, diabetic tractional retinal detachment) with either preserved crystalline lens or previous cataract surgery (at least 3 months prior to PPV) will be recruited

Exclusion Criteria:

Patient with previous history of ocular trauma, co-existing glaucoma, co-existing anterior uveitis, complicated cataract surgery, IOL-related complications, previous vitreo-retinal surgery, visually significant cataract (necessitating combined phacoemulsification with PPV and SO) and significant corneal opacity will be excluded. If any significant post-PPV complication develops, patient will be excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
central anterior chamber depth | 1 week
  Mean change in central anterior chamber depth after PPV with SO tamponade.

SECONDARY OUTCOMES:
peripheral anterior chamber depth | 1 week
  Mean change in peripheral anterior chamber depth
anterior chamber angle | 1 week
  mean change in anterior chamber angle
anterior chamber angle entry area | 1 week
  mean change anterior chamber angle entry area